CLINICAL TRIAL: NCT03039361
Title: Equine Assisted Psychotherapy for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-547
Record Dates: First submitted 2017-01-11; First posted 2017-02-01 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: PostTraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Equine Assisted Psychotherapy (Experimental): 6 week Equine Assisted Psychotherapy program
  Interventions: Behavioral: Equine Assisted Psychotherapy
- Control (No Intervention): Standard of Care, Existing PTSD therapy

INTERVENTIONS:
Behavioral: Equine Assisted Psychotherapy — Therapist will use Equine Assisted Growth and Learning Association (EAGALA) modeled Equine Assisted Psychotherapy.
  Other Names: Equine Assisted Therapy
  Arms: Equine Assisted Psychotherapy

SUMMARY:
The purpose of this study is to assess the efficacy of Equine Assisted Psychotherapy on PTSD symptoms in veterans with PTSD as compared with existing care.

The investigators' hypothesis is: EAP Participants' will experience decreased PTSD symptoms following participation in a 6-week Equine Assisted Psychotherapy program.

DETAILED DESCRIPTION:
This study will employ a randomized, parallel group design with delayed intervention in the control group. Eligible participants will be randomly assigned using a random number generator. The PTSD Checklist (PCL) - Military (measuring PTSD symptoms) will be administered to each participant at week 0 and week 6. Permissions have been obtained for the use of the survey.

Surveys will be identified by randomized number only, to maintain confidentiality. Participants will be assigned a unique identifier. A list of participant's initials and their random assigned numbers will be kept in a locked secure file by the investigator. In this way the participants confidentially will be protected.

The participants assigned to the intervention group will complete the Equine Assisted Psychotherapy (EAP) program that will be performed at an Equine Assisted Growth and Learning Association (EAGALA) certified facility. The participants will be going through a 6 week program. The researcher will not be conducting the therapy. An EAGALA certified and licensed Occupational Therapist will be running the therapy as well as a professional Horse Handler for safety. In the event that a participant is in need of additional therapy as a result of this research, a psychotherapist will be on call. Participation will not include riding the horses. "The basis of the EAGALA Model is a belief that all clients have the best solutions for themselves when given the opportunity to discover them. Rather than instructing or directing solutions, [the instructor] allow [their] clients to experiment, problem-solve, take risks, employ creativity, and find their own solutions that work best for them. No horseback riding is involved. Instead, effective and deliberate techniques are utilized where the horses are metaphors in specific ground-based experiences." (http://www.eagala.org/Information/What_Is_EAGALA_Model) All horse based activities involve inherent risk. The facility and the horses that the participants will be using are used daily for Hippotherapy involving disabled individuals. All safety procedures and precautions outlined by the EAGALA certifications and the therapy facility will be strictly maintained. The participants may decline to do any of the therapy activities and or survey questions at any time. If the certified therapist senses a problem, they will stop the therapy and consult with a psychotherapist.

The participants assigned to the control group will have no intervention related to the research but may continue any preexisting therapy. They will be asked to not initiate any new therapy programs. The participants will be however given the option of delayed EAP after the completion of the 6 week program.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include war veterans with post-traumatic stress disorder, who have a PCL-M symptom score of ≥ 29 with an age between 18 and 75.

Exclusion Criteria:

* Adults unable to consent, individuals aged < 18 years, individuals receiving antipsychotic medication, individuals receiving glucocorticoid therapy, and/or pregnant women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in 17-item PCL-Military (PTSD Symptoms) | Baseline and 6 weeks
  A validated and widely used survey instrument to assess PTSD symptoms for the purposes of diagnosis, clinical assessment, and scientific inquiry. Scores range from 17 to 85 in severity, with anything over 29 as having PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Burge, MD, Principal Investigator — UNM Clinical Translational Science Center

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be provided in Lobo vault after finalization of the study.